CLINICAL TRIAL: NCT03233477
Title: Patient Registry of Posner-Schlossman Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Chun Zhang, Professor, Peking University
Other Study IDs: IRB00006761-2014166
Record Dates: First submitted 2017-07-22; First posted 2017-07-28 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Posner Schlossman Syndrome
Keywords: Posner Schlossman Syndrome; cytokine expression; cytomegalovirus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — serum, aqueous humor，iris，trabecular meshwork
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Posner-Schlossman Syndrome: Inclusion criteria：
  * Clinical diagnosis of Posner-Schlossman Syndrome
  * Able to communicate with doctor and understand this study
  Exclusion criteria:
  * Not be able to communicate with doctor and understand this study
  * One or more authorized investigators think he or she will suffer from any severe risks from the study
- cataract: Inclusion criteria：
  * Clinical diagnosis of age-related cataract
  * Prepare for cataract operation
  * Open angle and intraocular pressure is normally at anytime
  * No family history of glaucoma
  Exclusion criteria:
  * Patients above 65 years old
  * With Secondary ocular hypertension
  * Have the history of receiving any ophthalmologic operation or anti-viral therapy
  * With diabetes mellitus
  * With autoimmune disease
  * Be receiving any therapy that can influence the virus-infection state and biochemical characteristics of serum and aqueous humor, or have received such therapy before one month
- primary open-angle glaucoma: Inclusion criteria：
  * Both eyes involved
  * Open angle
  * Progressive glaucomatous optic neuropathy
  * Specific visual field loss of glaucoma
  * Intraocular pressure above the up limit of normal people
  Exclusion criteria:
  * Patients above 65 years old
  * With Secondary ocular hypertension
  * Have the history of receiving any ophthalmologic operation or anti-viral therapy
  * With diabetes mellitus
  * With autoimmune disease
  * Be receiving any therapy that can influence the virus-infection state and biochemical characteristics of serum and aqueous humor, or have received such therapy before one month

SUMMARY:
Posner-Schlossman syndrome, or glaucomatocyclitic crisis, is a condition characterized by recurrent, acute attacks of mild, nongranulomatous, anterior uveitis accompanied by markedly elevated intraocular pressure. Most of patients are the 20 to 50-year-old young adults, with unilateral eye involvement. PSS was originally deemed benign, but is now recognized as a relatively rare cause of chronic secondary glaucoma,especially in patients with recurrent episodes. This relatively rare disease is likely the result of the infections of a variety of organisms, and the bulk of literature supports the cytomegalovirus (CMV) as the leading cause.

This study is an observational study that does not interfere with the normal clinical diagnosis and treatment process. The investigators in this study focus on observing the clinical symptoms and outcome of PSS, analyzing the factors that affect the prognosis of PSS, studying the association of its pathogenesis with the psychological status and the behavioral types of PSS patients; exploring the relationship between infection (CMV, HSV, Hp) and PSS; and studying the changes of local and systemic cytokine expression and its significance in patients with PSS.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to take part in this study and sign informed consent by oneself or the patient's legal representative
* Clinical diagnosis of Posner-Schlossman Syndrome, age-related cataract, or primary open-angle glaucoma
* Live in Beijing, China or being able to visit the Peking University Third Hospital every year after the beginning of the study or whenever the disease relapses

Exclusion Criteria:

* Fit any exclusion criteria of the patient's group

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the patients that visit the Peking University Third Hospital from July 2014 to July 2019 and are diognosed as Posner-Schlossman Syndrome, age-related cataract, or primary open-angle glaucoma.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2014-07-31 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
demographic characteristics | up to 10 years
  age, sex, education level, systemic disease， mental state
visual acuity | up to 10 years
  uncorrected visual acuity and best corrected visual acuity
intraocular pressure | up to 10 years
  Goldmann
slit-lamp examination | up to 10 years
  anterior segment
fundus photograph | up to 10 years
  analysis the morphology of optic nerve head
OCT | up to 10 years
  zess
visual field | up to 10 years
  Humphrey visual field
blood serum | up to 10 years
  8ml
aqueous humor | up to 10 years
  0.2ml
tissue | in the operation
  iris and& or trabecular meshwork tissue abandoned in the anti-glaucoma operation

CONTACTS AND LOCATIONS:
Overall Officials: Chun Zhang, PHD，MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hosipital, Beijing, Beijing Municipality, China